CLINICAL TRIAL: NCT01566396
Title: Evaluation of Safety and Efficacy of the 3F Applicator (A3F) for Treatment of Facial Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pollogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC210117_F, rev. 01
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-05

CONDITIONS: Facial Wrinkles
Keywords: Fractional,; RF,; Wrinkles; Safety; Efficacy; treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A3F (Experimental): A3F, Fractional RF treatment
  Interventions: Device: A3F

INTERVENTIONS:
Device: A3F — A3F fractional RF treatments for facial wrinkles

SUMMARY:
The 3F Applicator (A3F) is indicated for use in dermatological procedures requiring ablation and resurfacing of the skin, and for the treatment of facial wrinkles. This study was designed in order to evaluate the safety and efficacy of the A3F for treatment of facial wrinkles.

DETAILED DESCRIPTION:
The need for cosmetic facial enhancement procedures with minimal down time and low risk has led to the development of methods for non-surgical skin rejuvenation. Various ablative lasers were developed, which remove the full skin surface in a controlled manner1,2. However, the prolonged recovery and the significant risks prompted the development of fractional lasers which ablate the skin in a fractional manner, leaving untreated areas to improve healing process3. In the past few years, fractional RF systems have been introduced that enable controlled skin resurfacing accompanied with dermal collagen remodeling4,5,6. The new 3F Applicator (A3F, trade name TriFractional) from Pollogen™ is designed to enable skin resurfacing and treatment of wrinkles using radiofrequency energy.

The 3F Applicator (A3F) is indicated for use in dermatological procedures requiring ablation and resurfacing of the skin, and for the treatment of facial wrinkles. This study was designed in order to evaluate the safety and efficacy of the A3F for treatment of facial wrinkles.

ELIGIBILITY:
Inclusion Criteria:

1. Subject read, understood and signed the Consent Form
2. Healthy female/male aged 35 65 years,
3. Fitzpatrick wrinkle classification score 3 and above
4. Fitzpatrick skin type 2-5
5. Subject is capable of reading, understanding and following instructions of the procedure to be applied.
6. Subject is able and willing to comply with the treatment and follow-up schedule.

Exclusion Criteria:

1. Subject has a pacemaker or internal defibrillator, implanted neurostimulators or any other internal electric device or patient who had an implant in the past.
2. Subject has metal or other implants in the treatment area (Not including dental fillings, implants and crowns).
3. Subject has current or history of cancer, especially skin cancer or premalignant moles or is undergoing any form of treatment for active cancer.
4. Subject has severe concurrent conditions such as epilepsy, lupus or cardiac disorders.
5. Subject has poorly controlled endocrine disorders such as diabetes.
6. Subject is female who is pregnant, lactating, or plans to become pregnant during the study period or had given birth less than 6 months ago.
7. Subject has an impaired immune system due to immunosuppressive diseases such as HIV or AIDS, or use of immunosuppressive medications.
8. Subject has a condition that could be negatively affected by heat, including any history of diseases stimulated by heat, such as recurrent Herpes Simplex (in the treatment area).
9. Subject has diminished or exaggerated perception of temperature changes.
10. Subject has significant concurrent skin conditions affecting areas to be treated such as sores, hemorrhages or risk of hemorrhages, septic conditions, psoriasis, eczema and rash as well as very dry and fragile skin.
11. Subject has history of collagen disorders, keloid formation and abnormal wound healing.
12. Subject has had previous invasive/ablative procedures in the areas to be treated within 3 months prior to initial treatment or plans on such treatment during the course of the study, or before complete healing has occurred.
13. Subject has had Botox injections in the treatment area within 6 months prior to initial treatment
14. Subject has had natural fillers within 9 months prior to initial treatment
15. Subject has synthetic fillers, injected chemical substance or gold/plastic threads in the treatment area.
16. Subject takes or has taken medications, herbal preparations, food supplements or vitamins that might cause fragile skin or impaired skin healing such as prolonged steroid regime, tetracyclines, or St. John's Wort for the last 3 months.
17. Subject has used oral isotretinoin (Accutane or Roaccutan) within 6 months prior to study enrollment or plans use during the course of the study.
18. Subject has history of bleeding coagulopathies or use of anticoagulants.
19. Use of non-steroidal anti inflammatory drugs (NSAIDS, e.g. ibuprofen containing agents) one week before and after each treatment session prior to treatment
20. Tattoo or permanent makeup in the treated area
21. Subject has burned, blistered, irritated, or sensitive skin due to excessive fresh tanning in areas to be treated or is unlikely to refrain from excessive tanning during the study.
22. Concurrent participation in any other study.
23. Subject has mental disorders that in the opinion of the Investigator would be interfere with ability to comply with the study requirements.
24. Subject is allergic to the topical anesthetic used in this study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the 3F Applicator (A3F) for treatment of facial wrinkles. | 6 months
  The safety of using the 3F Applicator (A3F) for treatment of facial wrinkles a will be established by physician's assessment/observation of adverse events. AEs will be tabulated by severity and relation to treatment.

SECONDARY OUTCOMES:
To evaluate the efficacy of the 3F Applicator (A3F) for treatment of facial wrinkles. | 6 months
  Efficacy of using the 3F Applicator (A3F) for treatment of facial wrinkles will be established by level of wrinkle reduction. The treated area will be photographed, using high-resolution macro photography prior to the treatments and at the follow up visits. The pre - and post-treatment photographs will be compared and scored by two independent uninvolved physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Mira Barki, PhD, Study Director — Pollogen Ltd.
Locations (2):
- United States (2):
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Research Across America, Plano, Texas